CLINICAL TRIAL: NCT06158360
Title: A Prospective Multi-centered Observational Study on Postoperative Symptoms After Thyroidectomy (POS-T) in Patients with Thyroid Cancer
Brief Title: An Observational Study on Postoperative Symptoms After Thyroidectomy (POS-T)
Status: Recruiting | Type: Observational
Sponsor: Ilsan Cha hospital (Other)
Responsible Party: Principal Investigator, Jee Young Lee, Assistant professor, CHA University
Other Study IDs: ICICC-OS-23-01
Record Dates: First submitted 2023-11-06; First posted 2023-12-06 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Thyroid Cancer
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Axiom Asia Precision Medicine Research Array (PMRA) chip
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This observational study aimed to evaluate the safety and efficacy of postoperative management in patients with thyroid cancer who received subtotal or total thyroidectomy.

DETAILED DESCRIPTION:
1. Characteristic analysis of improvement in quality of life and symptoms after surgery in cancer patients
2. Multifaceted symptom evaluation of cancer patients visiting medical institutions
3. Evaluation of effectiveness and safety of treatment for postoperative symptoms in thyroid cancer patients
4. Analysis of the effectiveness and prognosis of cancer-related treatment for each patient with cancer
5. Analysis of prognostic factors for disease-free survival and overall survival of cancer patients

Among adult men and women aged 19 years or older who have been diagnosed with thyroid cancer, who have undergone partial or total thyroidectomy and visited the hospital for postoperative management, the characteristics of the visiting patient, quality of life, characteristics of cancer-related symptoms, and treatment effectiveness, We intend to conduct a prospective observational study to evaluate safety and its relationship with prognosis. In addition, we aim to form the basis for follow-up research through the establishment of an Oriental medicine cancer cohort and database.

ELIGIBILITY:
Inclusion Criteria:

* 19 years of age or older
* Those who have been confirmed to have a malignant tumor of the thyroid gland by biopsy or imaging
* Subjects who have undergone partial thyroidectomy or total resection within 1 month
* Those who have agreed to the implementation of Chinese medicine treatment
* The Eastern Cooperative Oncology Group(ECOG) performance status 0-3
* Those who understand the content of the study and agree to participate in the study

Exclusion Criteria:

* ○ When it is judged that other diseases other than cancer (dementia, cerebrovascular disease, severe organ failure, etc.) may have a significant effect on the decline of physical function

  * When it is judged that the life expectancy is less than 3 months and sufficient follow-up cannot be carried out
  * When emergency or major surgery or surgical intervention is required that takes precedence over postoperative treatment
  * Pregnant and lactating women
  * Other researchers who are judged to be unsuitable for research

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have been diagnosed with thyroid cancer (KCD C73) according to the ICD-10 International Classification of Diseases and have been recommended for postoperative management treatment by a physician or acupuncturist
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
THYCA-QoL score at the time of discharge (1w) of hospitalization performed for postoperative management purposes | At the end of week 1(each cycle is 7days)
  The THYCA-QoL is a health-related quality of life questionnaire developed for thyroid cancer and thyroid cancer survivors using methodologically proven standard guidelines and validated questionnaires to improve symptoms, treatment, follow-up and disease experience in thyThe THYCA-QoL is a health-related quality of life questionnaire developed for thyroid cancer and thyroid cancer survivors using methodologically proven standard guidelines and validated questionnaires to improve symptoms, treatment, follow-up and disease experience in thyroid cancer survivors. roid cancer survivors.

SECONDARY OUTCOMES:
Change in THYCA-QoL over time series | At the end of Day 1, week 1, week 2, 1 month, 2 month, 3 month, 4 month, 6 month, 12 month
  The THYCA-QoL is a health-related quality of life questionnaire developed for thyroid cancer and thyroid cancer survivors using methodologically proven standard guidelines and validated questionnaires to improve symptoms, treatment, follow-up and disease experience in thyThe THYCA-QoL is a health-related quality of life questionnaire developed for thyroid cancer and thyroid cancer survivors using methodologically proven standard guidelines and validated questionnaires to improve symptoms, treatment, follow-up and disease experience in thyroid cancer survivors. roid cancer survivors.
EORTC-QLQ-C30 | At the end of Day 1, week 1, week 2, 1 month, 2 month, 3 month, 4 month, 6 month, 12 month
  It is a health-related questionnaire for cancer patients. It consists of 3 subdomains: overall quality of life, functional area, and symptom domain, a total of 30 items.
BCQ | At the end of Day 1, week 1, week 2
  It is a dialectic tool that divides the physiological and pathological conditions and symptoms of the human body into three dialectics: concession, yinhe, and word-body, and identifies the deteriorated condition of the human body.
CHPIQ | At the end of Day 1, week 1, week 2
  It is a key diagnostic technology that plays a decisive role in the selection of prescriptions in traditional Chinese medicine, and it is a symptom-based cold and heat pattern identification questionnaire that has been recognized for its reliability and validity. CHPIQ).
MDASI-Core | At the end of Day 1, week 1, week 2, 1 month, 2 month, 3 month, 4 month, 6 month, 12 month
  The MDASI-core is a 19-item questionnaire that identifies pain, fatigue, nausea, vomiting, insomnia, shortness of breath, cognitive function, anorexia and dysthymia on a 10-point scale.
Oral epithelial cell-based whole genome analysis | Day 1
  The Asia PMRA chip contains more than 300 cancer-related common variants and 2,600 rare variants as well as 2,600 pharmacogenomic-related variants, including more than 300 cancer-related common variants and 2,600 rare variants contained in the ClinVar (> 43,000 markers) or GWAS Catalog (> 23,400 markers), which are databases for diseases and various traits.
overall survival | At the end of Day 1, week 1, week 2, 1 month, 2 month, 3 month, 4 month, 6 month, 12 month
  To investigate the overall survival of study subjects enrolled in the study and cancer-related deaths, from the time of initiation of cancer-related TCM treatment to death.
Adverse events | At the end of Day 1, week 1, week 2, 1 month, 2 month, 3 month, 4 month, 6 month, 12 month
  CTCAE ver. To investigate the types and incidence of adverse events in accordance with 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Jee Youg Lee, Principal Investigator — Ilsan Cha hospital
Locations (3):
- South Korea (3):
  - Bundang Cha Hospital, Gyeonggi-do
  - Ilsan Cha Hospital, Gyeonggi-do
  - Gangnam Cha Hospital, Seoul